CLINICAL TRIAL: NCT03127319
Title: A Study of Apatinib Plus Docetaxel for Treatment of Advanced Non-squamous Non-small Cell Lung Cancer With Bone Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Hebei University (Other)
Responsible Party: Principal Investigator, Aimin Zang, Director of oncology, Affiliated Hospital of Hebei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHHU-2017AMZ01
Record Dates: First submitted 2016-12-30; First posted 2017-04-25 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-01

CONDITIONS: Non-squamous Non-small Cell Lung Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- apatinib and docetaxel zoledronic (Experimental): apatinib 500mg qd po; docetaxel 60mg/m² iv q3w; zoledronic 4mg iv>15min q4w until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: apatinib docetaxel zoledronic
- docetaxel zoledronic (Active Comparator): docetaxel 60mg/m² iv q3w;zoledronic 4mg iv>15min q4w until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: docetaxel zoledronic

INTERVENTIONS:
Drug: apatinib docetaxel zoledronic — apatinib 500 mg qd p.o.docetaxel 60mg/m² iv q3w;zoledronic 4mg iv>15min q4w until disease progression or intolerable toxicity or patients withdrawal of consent
  Arms: apatinib and docetaxel zoledronic
Drug: docetaxel zoledronic — docetaxel 60mg/m² iv q3w;zoledronic 4mg iv>15min q4w until disease progression or intolerable toxicity or patients withdrawal of consent
  Arms: docetaxel zoledronic

SUMMARY:
The purpose of this study is to assess the efficacy and safety of patients who receive apatinib plus docetaxel and zoledronic versus docetaxel and zoledronic alone as second line treatment for advanced non-squamous non-small cell lung cancer with bone metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 to 75 years old (man or female)
2. Pathologically diagnosed with metastatic or recurrent non-squamous non-small cell lung cancer
3. Patients with at least one evaluate lesions of the lung and bone metastases.(measuring≥10mm on spiral CT scan, satisfying the criteria in RECIST1.1 and WHO)
4. Refractory or failure of prior therapy
5. Life expectancy greater than or equal to 3 months
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
7. Major organ function has to meet the following criteria:

   * For results of blood routine test (without blood transfusion within 14 days)

     1. HB≥90g/L
     2. ANC≥1.5×109/L
     3. PLT≥180×109/L
   * For results of blood biochemical test：

     1. TBIL<1.5×ULN；
     2. ALT and AST<2.5×ULN, but< 5×ULN if the transferase elevation is due to liver metastases；
     3. Serum creatinine ≤1.25×ULN , or calculated creatinine clearance>45 ml/min(per the Cockcroft-Gault formula);
8. Women of childbearing age must have contraceptive measures or have test pregnancy (serum or urine) enroll the study before 7 days, and the results must be negative, and take the methods of contraception during the test and the last to have drugs after 8 weeks. Men must be contraception or has sterilization surgery during the test and the last to have drugs after 8 weeks;
9. Participants were willing to join in this study, and written informed consent, good adherence, cooperate with the follow-up.

Exclusion Criteria:

1. Allergic to apatinib and docetaxel;
2. Have high blood pressure and antihypertensive drug treatment can not control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg), with class Ⅱ and above coronary heart disease, arrhythmia (including QTc lengthened men > 450 ms, women > 470 ms) and class Ⅲ-Ⅳ cardiac insufficiency;
3. A variety of factors influencing oral drugs (such as unable to swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc.).
4. Patients with tendency of gastrointestinal bleeding, including the following: a local active ulcerative lesions, and defecate occult blood (+ +); Has melena and hematemesis in two months; For defecate occult blood (+) and primary lesions without surgical removal of the stomach tumor, requirement of gastroscopy, such as ulcer type of gastric cancer, and researchers think that may be gastrointestinal hemorrhage;
5. Coagulant function abnormality (INR > 1.5 ULN, APTT > 1.5 ULN), with bleeding tendency.
6. Patients with symptoms of central nervous system metastasis.
7. Pregnant or lactating women.
8. history of psychiatric drugs abuse and can't quit or patients with mental disorders.
9. Less than 4 weeks from the last clinical trial.
10. The researchers think inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-03 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | evaluation per 2 cycles (6 weeks)

SECONDARY OUTCOMES:
Overall survival | evaluation per 2 cycles (6 weeks)
DCR (Disease control rate) | evaluation per 2 cycles (6 weeks)
ORR (Objective response rate) | evaluation per 2 cycles (6 weeks)
SREs（Skeletal-related events） | evaluation per 2 cycles (6 weeks)
  measured pain, a fracture, the need for bone radiation or surgical therapy, spinal cord compression, or hypercalcemia
Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 | evaluation per 2 cycles (6 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Hebei university, Baoding, Hebei, China